CLINICAL TRIAL: NCT06128863
Title: Phase II, Single-arm Clinical Trial Evaluating Efficacy and Safety of Pembrolizumab in Combination With a Soluble LAG-3 Protein, Eftilagimod Alpha, and Radiotherapy in Neoadjuvant Treatment of Patients With Soft Tissue Sarcomas (EFTISARC-NEO)
Brief Title: Pembrolizumab in Combination With Eftilagimod Alpha and Radiotherapy in Neoadjuvant Treatment of Patients With Soft Tissue Sarcoma - EFTISARC-NEO Trial
Acronym: EFTISARC-NEO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Immutep S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFTISARC-NEO/NIO-0004; 2022-003845-36 (EudraCT Number)
Record Dates: First submitted 2023-10-28; First posted 2023-11-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-02

CONDITIONS: Neoadjuvant; Immunotherapy; Sarcoma,Soft Tissue; Radiation Therapy
Keywords: soft tissue sarcoma; immunotherapy
MeSH Terms: conditions — Sarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other): Systemic therapy with pembrolizumab and eftilagimod alfa is given concurrently with radiotherapy.
  Surgery is scheduled 5-6 weeks after completion of radiotherapy.
  Interventions: Drug: Pembrolizumab, Eftilagimod alfa

INTERVENTIONS:
Drug: Pembrolizumab, Eftilagimod alfa — Eftilagimod alfa 20 mg s.c. every 2 weeks (5 doses), Pembrolizumab 200 mg i.v. every 3 weeks (3 cycles), Radiotherapy 50 Gy (25 x 2 Gy)
  Other Names: Keytruda; Eftilagimod alfa; Efti

SUMMARY:
This is a phase II single-arm single-stage study evaluating efficacy and safety of pembrolizumab in combination with a soluble LAG-3 protein, eftilagimod alfa (Efti) and radiotherapy in neoadjuvant treatment of patients with soft tissue sarcomas. This study will determine the pathologic response rate (defined as percentage of tumor hyalinization/fibrosis) to the combination treatment.

DETAILED DESCRIPTION:
Systemic therapy with pembrolizumab and eftilagimod alfa and radiotherapy are administered concurrently. Systemic treatment lasts for 9 weeks (study week 1-9). Radiation therapy lasts for 5 weeks (5 days per week) in weeks 2-6. Surgery takes place 5-6 weeks after completion of radiation therapy (week 11-12). Any adjuvant treatment (chemotherapy, immunotherapy, radiation therapy) after surgical treatment is not allowed. Patients will be then followed up regularly for a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary or locally recurrent deep-seated extremities, girdles and/or superficial trunk (thoracic or abdominal wall) soft tissue sarcoma
* Grade 2 or 3 tumors according to Fédération Nationale des Centres de Lutte contre le Cancer (FNCLCC);
* Size of the primary tumor >5 cm at instrumental staging (CT, MRI), or locally recurrent of any size;
* Measurable disease based on RECIST 1.1;
* Non-metastatic disease;

Exclusion Criteria:

* Ewing sarcoma, Alveolar and embryonal rhabdomyosarcoma
* Previous treatment with eftilagimod alfa, anti-PD-1 or anti-PD-L1;
* Prior radiotherapy to tumor-involved sites;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic response | At the time of definitive surgical treatment
  The primary efficacy endpoint is a percent tumor hyalinization as a marker of response to treatment assessed at the time of surgical resection.

SECONDARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | All adverse events will be documented from the enrolment of the first patient until 100 days after the surgical treatment of the last patient (2 years).
  Safety analyses will include all patients who received at least one dose of study drug. Safety will be assessed through summaries of adverse events, changes in laboratory test results, changes in vital signs.
  Verbatim description of adverse events will be summarized and graded according to International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. In addition, serious adverse events, severe adverse events (Grades 3, 4, and 5), and adverse events leading to study drug discontinuation or interruption will be summarized accordingly.
Number of participants completing neoadjuvant therapy | 2 years
  Number of patients completing neoadjuvant treatment and having a curative surgery according to the protocol
Disease-free survival (DFS) | From the date of curative surgery to the date of first recurrence or death (whatever the cause), whichever occurs first
  Disease-free survival (DFS) is defined as the time from between the date of curative surgery and the date of disease recurrence defined as clinically diagnosed or biopsy-confirmed recurrent sarcoma at a site of the primary tumor, development of nodal metastasis, locoregional recurrence or distant metastases confirmed by imaging or clinical examination, or death without documented recurrence
Local recurrence-free survival (LRFS) | From the date of curative surgery to the date of first local recurrence or date of death (whatever the cause), whichever occurs first
  Local recurrence-free survival (LRFS) is defined as the time between the date of curative surgery and the date of local recurrence confirmed by imaging or clinical examination. Patients still alive and without signs of disease recurrence at the analysis cut-off date are censored at the last date known to be alive.
Distant metastasis-free survival (DMFS) | From the date of curative surgery to the date of first distant metastasis or date of death (whatever the cause), whichever occurs first
  Distant metastasis-free survival (DMFS) is defined as the time between the date of curative surgery to the date of diagnosis of distant metastases confirmed by imaging or clinical examination. Patients still alive and without signs of distant metastases at the analysis cut-off date are censored at the last date known to be alive.
Overall survival (OS) | From the date of curative surgery up to the date of death or the last date the participant was known to be alive
  Overall survival (OS) is defined as the time between the date of curative surgery and the date of death from any cause. For those without documentation of death, OS will be censored on the last date the participant was known to be alive.
Response rate | From the date of the first dose of treatment to the date of curative surgery
  Radiologic Response To Neoadjuvant Treatment using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Kozak, Principal Investigator — Maria Sklodowska-Curie National Research Institute of Oncology
Locations (1):
- Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland